CLINICAL TRIAL: NCT07102888
Title: A Phase II Clinical Study to Evaluate the Safety and Pharmacokinetics of Topical RSS0393 Ointment in Children and Adolescents With Plaque Psoriasis
Brief Title: A Clinical Study to Evaluate the Safety and Pharmacokinetics of Topical RSS0393 Ointment in Children and Adolescents With Plaque Psoriasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSS0393Oint-203
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Plaque Psoriasis in Children; Plaque Psoriasis in Adolescents

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RSS0393 Ointment Group (Experimental)
  Interventions: Drug: RSS0393 Ointment

INTERVENTIONS:
Drug: RSS0393 Ointment — RSS0393 ointment.

SUMMARY:
This study is to evaluate the safety, tolerability, pharmacokinetics and efficacy of RSS0393 topical ointment in the treatment of plaque psoriasis in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 6 years old and < 18 years old at screening.
2. History of plaque psoriasis ≥ 3 months.
3. The subjects and their parents or legal guardians voluntarily signed informed consent before any study-related procedures began.

Exclusion Criteria:

1. Diagnosis of psoriasis other than plaque at screening.
2. Subjects have other skin diseases or conditions that may affect the evaluation of the relevant endpoints of this study.
3. Subjects with any other persistent active autoimmune disease.
4. Subjects who have received topical medication for psoriasis within 14 days before baseline, or systemic medication or phototherapy for psoriasis within 28 days before baseline, or biological agents for psoriasis within a specified time before baseline.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs). | About 4 weeks.

SECONDARY OUTCOMES:
The trough concentration of RSS0393. | About 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided